CLINICAL TRIAL: NCT05469971
Title: Contribution of KIR Genes on the Genetic Predisposition to Non-Celiac Wheat Sensitivity
Brief Title: KIR Genes and Non-Celiac Wheat Sensitivity
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, Associate Professor, University of Palermo
Other Study IDs: ACPM29
Record Dates: First submitted 2022-07-11; First posted 2022-07-22 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Non-celiac Wheat Sensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — A venous blood sample will be taken for each patient (1 dry tube and 1 EDTA tube). Blood samples will be stored at -80°C and subsequently used for DNA extraction and KIR genotyping by KIR SSO Genotyping Test (One Lambda, Thermo Fisher, Monza, Italy).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NCWS patients: The researchers will enrol NCWS, presenting with IBS and/or dyspepsia-like symptoms, according to the Rome IV criteria (20). These patients were diagnosed by DBPC wheat challenge between January 2010 and June 2022 in three tertiary centers for "gluten-related disorders" (Department of Internal Medicine, University Hospital of Palermo, Italy; Department of Internal Medicine, "Cervello" Hospital of Palermo, Italy, and Department of Internal Medicine, Hospital of Sciacca, Agrigento, Italy.
  Interventions: Genetic: KIR genotyping
- Celiac disease: The researchers will enrol CD patients diagnosed between January 2010 and June 2022 in three tertiary centers for "gluten-related disorders" (Department of Internal Medicine, University Hospital of Palermo, Italy; Department of Internal Medicine, "Cervello" Hospital of Palermo, Italy, and Department of Internal Medicine, Hospital of Sciacca, Agrigento, Italy.
  Interventions: Genetic: KIR genotyping
- Blood donors: The researchers will enroll blood donors from the Transfusion Centre of the University Hospital of Palermo, Italy.
  Interventions: Genetic: KIR genotyping

INTERVENTIONS:
Genetic: KIR genotyping — DNA extraction and KIR genotyping by KIR SSO Genotyping Test (One Lambda, Thermo Fisher, Monza, Italy).

SUMMARY:
Non-celiac gluten sensitivity (NCGS) is a condition characterized by gastrointestinal and extraintestinal symptoms which are triggered by gluten ingestion in the absence of celiac disease (CD) and wheat allergy. In the last years studies suggested that wheat components other than gluten can be responsible of symptom's triggering, thus the term "non-celiac wheat sensitivity" (NCWS) has been proposed as a more appropriate label. To date, different pathogenetic mechanisms have been proposed, but no conclusive data have been reported; among these, some study groups a possible role of innate immunity and of Natural Killer (NK) cells. KIR (Killer Immunoglobulin-like Receptors) regulate the activation of NK cells through their interaction with Human Leucocyte Antigens (HLA). Both KIR and HLA loci are highly polymorphic, and, in the case of KIR, two main haplotypes have been identified: A and B. Haplotype A is the simplest and correlates mainly with NK inhibition, while haplotype B has a variable number of genes, most of which activate NK cells. The investigators hypothesis is that the genetic variants of KIR, which define the haplotype "inhibitor" or "activator", can affect the development and the course of NCWS too. Thus, the researchers aimed to:1. Identify putative KIR genetic variants in NCWS patients (50 subjects) respect to celiac disease patients (50 subjects) and blood donors (50 subjects); 2. Evaluate the possible association of KIR genetic variants with specific clinical manifestations of patients with NCWS.

DETAILED DESCRIPTION:
Non-celiac gluten sensitivity (NCGS) is a condition characterized by gastrointestinal and extraintestinal symptoms which are triggered by gluten ingestion in the absence of celiac disease (CD) and wheat allergy. Despite the great interest in NCGS, much remains unknown about its pathogenesis. Some studies seem to suggest that wheat components other than gluten (i.e. amylase/trypsin inhibitors, ATIs) can be responsible of symptom's triggering, and therefore the term "non-celiac wheat sensitivity" (NCWS) has been proposed as a more appropriate label. NCWS pathogenesis has been attributed to very different mechanisms: innate or adaptive immunity, incomplete digestion and/or absorption of fermentable oligosaccharides and disaccharides, monosaccharides, and polyols, and, finally, psychological effect. Although NCWS might be considered in its clinical features like CD, to date, no data are available about genes that confer a higher genetic predisposition to the disease. It is known that, in contrast to CD, patients with NCWS do not have a characteristic Human Leucocyte Antigens (HLA) genotype/phenotype, even if HLA DQ2/DQ8 alleles are present in 40-50% of these patients, a value higher than that of the general population (30%). Many studies ascertained the importance of innate immunity and of Natural Killer (NK) cells in the pathogenesis of NCWS. KIRs (Killer Immunoglobulin-like Receptors) regulate the activation of NK cells through their interaction with HLA. Both KIR and HLA loci are highly polymorphic, and, in the case of KIR, two main haplotypes have been identified: A and B. Haplotype A is the simplest and correlates mainly with NK inhibition, while haplotype B has a variable number of genes, most of which activate NK cells. More in general, several studies have shown that haplotypes containing predominantly activator genes confer protection against viral infections and susceptibility to the development of autoimmune and neoplastic diseases. In the context of CD, NK cells are one of the main components of innate immunity and are involved in the destruction of epithelial cells and their cytotoxic activity is closely related to the function of KIRs. The investigators hypothesis is that the genetic variants of KIR, which define the haplotype "inhibitor" or "activator", can affect the development and the course of NCWS too. Thus, the researchers aimed to: 1. Identify putative KIR genetic variants in NCWS patients (50 subjects) respect to celiac disease patients (50 subjects) and blood donors (50 subjects); 2. Evaluate the possible association of KIR genetic variants with specific clinical manifestations of patients with NCWS.

ELIGIBILITY:
1. Inclusion Criteria for NCWS patients

   * age >18 and <65 years
   * subjects with gluten/wheat-dependent symptoms, both intestinal and extra-intestinal
   * negativity of anti-deamidated gliadin protein (DGP) immunoglobulins (Ig) class A (IgA) and IgG, anti-tissue transglutaminase (tTG) IgA and IgG, Endomysium antibody (EMA)
   * absence of villous atrophy at the duodenal level, documented in all patients with HLA DQ2 and/or DQ8 (therefore, regardless of the negativity of CD-specific serum antibodies), evaluated when patients had a minimum intake of 100 grams of pasta and/or bread a day, for at least 45 days
   * absence of wheat allergy (negative prick-test and/or specific serum IgE assay for wheat, gluten and gliadin)
   * resolution of symptoms with a strict standard elimination diet, i.e., "oligoantigenic" (without wheat, cow's milk, egg, tomato and chocolate, and other foods self-reported by the patient as causing symptoms), for at least 4 weeks, followed by the reappearance of the same after a Double-Blind Placebo-Controlled Challenge (DBPCC) with gluten/wheat
   * complete medical records
   * duration of follow-up greater than 12 months after initial diagnosis and at least 2 outpatient visits during the follow-up period.
2. Exclusion Criteria for NCWS patients

   * age <18 and >65 years
   * alcohol and/or drug abuse
   * self-exclusion of gluten/wheat from the diet and refusal to reintroduce it, for diagnostic purposes, before entering the study
   * treatment with steroids and/or non-steroidal anti-inflammatory drugs (NSAIDs) in the 2 weeks prior to performing duodenal biopsies
   * positivity of EMA in the culture medium of duodenal biopsies, even in the presence of a normal villus/crypt ratio in the duodenal mucosa
   * incomplete medical records
   * lack of clinical follow-up of at least 12 months from diagnosis
   * pregnancy
   * diagnosis of chronic inflammatory bowel disease or other organic pathology affecting the digestive system, diseases of the nervous system, major psychiatric disorders, infectious diseases, immunological deficits, and impairments that limit physical activity.
3. Criteria for inclusion of patients with CD

   * age >18 and <65 years
   * subjects with gluten/wheat-dependent symptoms, both intestinal and extraintestinal, who meet the diagnostic criteria of CD reported in the current guidelines ("four out of five rule"): 1) typical intestinal and extraintestinal signs and symptoms of CD; 2) antibody positivity (both immunoglobulin (Ig) A class anti-tTG and EMA in IgA-sufficient or IgG class anti-tTG and EMA in IgA-deficient subjects); 3) HLA-DQ2 and/or -DQ8 positivity; 4) intestinal damage (demonstrated by histology on duodenal biopsies according to the Marsh classification); 5) clinical response to gluten-free diet (GFD) (e.g., resolution of intestinal and/or extra-intestinal symptoms).
4. Exclusion criteria for patients with CD

   * age <18 and >65 years
   * alcohol and/or drug abuse
   * incomplete medical records
   * lack of clinical follow-up of at least 12 months from diagnosis
   * pregnancy
   * diagnosis of chronic inflammatory bowel disease or other organic pathology affecting the digestive system, diseases of the nervous system, major psychiatric disorders, infectious diseases, immunological deficits and impairments that limit physical activity.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 50 NCWS patients, 50 CD patients, and 50 healthy blood donors.
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
KIR genetic variants in NCWS patients respect to CD patients and blood donors | Through study completion, an average of 1 year
  Evaluation of the presence and prevalence of KIR genetic variants (haplotype A or B) in NCWS patients respect to CD patients and blood donors.
Association between KIR genetic variants and clinical manifestation of NCWS patients | Through study completion, an average of 1 year
  Association between KIR genetic variants and the clinical symptoms (irritable bowel syndrome-like, functional dyspepsia-like, and extraintestinal) of NCWS patients.
Association between KIR genetic variants and associated autoimmune diseases of NCWS patients | Through study completion, an average of 1 year
  Association between KIR genetic variants and the associated autoimmune diseases (e.g., autoimmune thyroiditis) of NCWS patients.
Association between KIR genetic variants and coexistent other food allergies/intolerances of NCWS patients | Through study completion, an average of 1 year
  Association between KIR genetic variants and the coexistent other food allergies/intolerances (e.g., self-reported milk intolerance) of NCWS patients.
Association between KIR genetic variants and HLA DQ2-DQ8 genotypes of NCWS patients. | Through study completion, an average of 1 year
  Association between KIR genetic variants and the HLA DQ2-DQ8 genotypes of NCWS patients.
Association between KIR genetic variants and duodenal histology of NCWS patients. | Through study completion, an average of 1 year
  Association between KIR genetic variants and the duodenal histology (i.e., Marsh-Oberuber classification) of NCWS patients.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, MD, Study Chair — Department of Internal Medicine, "Cervello" Hospital of Palermo, Italy; Marcello Ciaccio, MD, Study Director — Institute of Clinical Biochemistry, University of Palermo, Italy
Locations (4):
- Italy (4):
  - Department of Internal Medicine, Giovanni Paolo II Hospital of Sciacca, Sciacca, Agrigento
  - Internal Medicine Division of the "Cervello-Villa Sofia" Hospital, Palermo, PA
  - Department of Biomedicine, Neurosciences and Advanced Diagnostics, Institute of Clinical Biochemistry, Clinical Molecular Medicine and Clinical Laboratory Medicine, University of Palermo, Palermo
  - Department of Internal Medicine, University Hospital of Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carroccio A, Soresi M, Chiavetta M, La Blasca F, Compagnoni S, Giuliano A, Fayer F, Mandreucci F, Castellucci D, Seidita A, Affronti A, Florena AM, Mansueto P. Frequency and Clinical Aspects of Neurological and Psychiatric Symptoms in Patients with Non-Celiac Wheat Sensitivity. Nutrients. 2021 Jun 8;13(6):1971. doi: 10.3390/nu13061971. PMID 34201313
- [Result] Mansueto P, Di Liberto D, Fayer F, Soresi M, Geraci G, Giannone AG, Seidita A, D'Alcamo A, La Blasca F, Lo Pizzo M, Florena AM, Dieli F, Carroccio A. TNF-alpha, IL-17, and IL-22 production in the rectal mucosa of nonceliac wheat sensitivity patients: role of adaptive immunity. Am J Physiol Gastrointest Liver Physiol. 2020 Sep 1;319(3):G281-G288. doi: 10.1152/ajpgi.00104.2020. Epub 2020 Jul 13. PMID 32658621
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Non-celiac gluten sensitivity: literature review. J Am Coll Nutr. 2014;33(1):39-54. doi: 10.1080/07315724.2014.869996. PMID 24533607
- [Result] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366
- [Result] Santin I, Castellanos-Rubio A, Perez de Nanclares G, Vitoria JC, Castano L, Bilbao JR. Association of KIR2DL5B gene with celiac disease supports the susceptibility locus on 19q13.4. Genes Immun. 2007 Mar;8(2):171-6. doi: 10.1038/sj.gene.6364367. Epub 2007 Jan 11. PMID 17215859
- [Result] Fernandez-Jimenez N, Santin I, Irastorza I, Plaza-Izurieta L, Castellanos-Rubio A, Vitoria JC, Bilbao JR. Upregulation of KIR3DL1 gene expression in intestinal mucosa in active celiac disease. Hum Immunol. 2011 Aug;72(8):617-20. doi: 10.1016/j.humimm.2011.04.008. Epub 2011 May 13. PMID 21616111
- [Result] Caggiari L, Toffoli G, De Re V, Orzes N, Spina M, De Zorzi M, Maiero S, Cannizzaro R, Canzonieri V. KIR/HLA combination associated with the risk of complications in celiac disease. Int J Biol Markers. 2011 Oct-Dec;26(4):221-8. doi: 10.5301/JBM.2011.8903. PMID 22180175
- [Result] Akar HH, Patiroglu T, Sevinc E, Aslan D, Okdemir D, Kurtoglu S. Contribution of KIR genes, HLA class I ligands, and KIR/HLA class I ligand combinations on the genetic predisposition to celiac disease and coexisting celiac disease and type 1 diabetes mellitus. Rev Esp Enferm Dig. 2015 Sep;107(9):547-53. doi: 10.17235/reed.2015.3817/2015. PMID 26334461